CLINICAL TRIAL: NCT02327949
Title: Prospective Comparison Between W-Shaped Acetabular Angular Plate (WAAP) and Reconstruction Plate for the Treatment of Posterior Acetabular Wall Fracture
Brief Title: W-Shaped Acetabular Angular Plate (WAAP) Versus Reconstruction Plate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhiyong Hou, Deputy Director of Orthopaedic Center,MD, Hebei Medical University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HZY-0001
Record Dates: First submitted 2014-12-20; First posted 2014-12-31 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Fracture of Posterior Wall of Acetabulum
MeSH Terms: interventions — Mandibular Reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- WP group (Experimental): WP group:treated with W-Shaped Angular Plate
  Interventions: Device: W-Shaped Angular Plate
- RP group (Active Comparator): RP group:treated with Reconstruction Plate
  Interventions: Device: Reconstruction Plate

INTERVENTIONS:
Device: W-Shaped Angular Plate — Treatment of posterior wall fracture of the acetabulum with a W-Shaped Angular Plate
  Arms: WP group
Device: Reconstruction Plate — Treatment of posterior wall fracture of the acetabulum with a Reconstruction Plate
  Arms: RP group

SUMMARY:
The purpose of this study is to determine whether this new W-Shaped Angular Plate is more effective and more safe to operate than the traditional reconstruction plate in the treatment of the posterior wall fracture of acetabulum.

DETAILED DESCRIPTION:
The posterior acetabular wall fracture is one of the simpler acetabular fracture patterns and the most common type, accounting for approximately one quarter of all acetabular fractures. Most patients achieve excellent outcomes after anatomical reduction and rigid internal fixation with standard screws and buttress plates.However,it is well known that the reconstruction plate need remould in the surgery. So it does not only lead to the extension of operation time, but also cause poor attach of acetabular posterior wall. Moreover, the angulation of the screw placement for the holes of the reconstruction plate in the danger zone was determined with only caution. The intraoperative fluoroscopy was employed frequently to help determine the periacetabular screw location. If the operator lack of experience, intraarticular screw penetration and prolonged operative duration is inevitable. The investigators now introduce a new type of internal fixation device of acetabular posterior wall fracture that improve the shortcomings of existing technology.The plate itself can be thought to consist of three regions: the iliac region, the danger zone region, and the ischial tuberosity region. The organization of these regions causes the plate to resemble the English alphabet letter ''W''.The contour and zygomorphy of the W-shaped plate matched the surface of the posterior column of the acetabulum. There are two rows of drill holes in the danger zone region. A special safe-angled drilling guide was used to assist in the operation. A retrospective study has been indicated that this kind of new plate produce good results. This device may help to avoid intraarticular screw penetration and reduce operative duration and blood loss. The device further provides a stable fixation of the posterior wall that is amenable to early range of motion and weight bearing postoperatively, and results in a good clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older(with no upper age limit)
* Sustained a posterior acetabular wall fracture(ASIF/OTA classification 62-A1)
* Operation was performed within 14 days after the fracture occurring

Exclusion Criteria:

* Presented with a pathologic acetabular fracture
* Neuropathic arthropathy,dementia and other disease processes which made postoperative compliance unreliable
* Refused to participate
* Patients who were unable to walk before injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Reduction quality of fracture | Six months
  Based on the radiographic grade criteria developed by Matta

SECONDARY OUTCOMES:
Surgical details | Intraoperative
  Operative duration,Fluoroscopy time,Blood loss, Blood transfusion,Any possible intraoperative complications
Early postoperative complications | One month
  Deep vein thrombosis (DVT), Skin necrosis, Infection, Loss of reduction, Arthritis,Death
Late postoperative complications | One year
  Heterotopic ossification, Chondrolysis, Avascular necrosis,Posttraumatic arthrosis
Evaluation of Clinical outcome | One year
  According to a modified Merle d'Aubigne and Postel score

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Hou, MD, Study Chair — Hebei Medical University Third Hospital; Shuai Shang, MM, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China